CLINICAL TRIAL: NCT04402892
Title: SARS-CoV-2 Specific Memory B and T- CD4+ Cells
Brief Title: COVID-19: SARS-CoV-2 Specific Memory B and T-CD4+ Cells
Acronym: MEMO-COV2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP200551
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; Immunity
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The recruitment of healed patients will be carried out via the Mondor and Bichat hospitals.
  After information and obtaining consent at D0 :
  * the patients will be taken from the departments of the participating centres (35 ml of blood, 5 LITHIUM HEPARINATE tubes).
  * Inpatients will be drawn from the wards of the participating centres (35 ml of blood, 5 LITHIUM HEPARINATE tubes).
  Inpatients will be drawn from the departments of the participating centres (35 ml of blood, 5 LITHIUM HEPARINATE tubes) at D21, then at D90 (3 months) for both groups of patients.
  Patients in both groups will be collected from the departments of the participating centres (35 ml of blood, 5 LITHIUM HEPARINATE tubes) at 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients hospitalized for SARS-CoV-2 (Active Comparator): Patients hospitalized for CoV-2-SARS will be sampled at inclusion (Day 0), at day 21, at 3 months and at 6 months .
  Interventions: Other: 35 ml blood, 5 tubes LITHIUM HEPARINATE at each time (hospitalized Patients )
- Patients who have recovered from CoV-2-SARS (Active Comparator): Patients who have recovered from CoV-2-SARS will be sampled at inclusion (Day 0), at 3 months and at 6 months .
  Interventions: Other: 35 ml blood, 5 tubes LITHIUM HEPARINATE at each time (cured Patients)

INTERVENTIONS:
Other: 35 ml blood, 5 tubes LITHIUM HEPARINATE at each time (hospitalized Patients ) — Patients hospitalized for CoV-2-SARS will be sampled at inclusion (Day 0), at day 21, at 3 months and at 6 months .
  Arms: Patients hospitalized for SARS-CoV-2
Other: 35 ml blood, 5 tubes LITHIUM HEPARINATE at each time (cured Patients) — Patients who have recovered from CoV-2-SARS will be sampled at inclusion (Day 0), at 3 months and at 6 months .
  Arms: Patients who have recovered from CoV-2-SARS

SUMMARY:
The current pandemic caused by the newly identified coronavirus responsible for COVID-19 is a major threat to our populations and societies.

Hypothesis/Objective The acquisition of protective immunity at the level of the individual, either through vaccination or natural resolution of the infection, progressively leads at the level of the population to the reduction of the fraction of the population that can be productively infected and transmit the virus, hence, leading to the diminution of the rate of transmission, a phenomenon called herd immunity. Herd immunity was proposed as a strategy to control the infection. However, it remains difficult to model group immunity given the limited knowledge of the interaction between the host immune system with the virus, whose capacity to evolve in face of a neutralizing response is also not known. It is therefore important to acquire a better knowledge of the immunological memory that ensures the resolution of COVID-19 after SARS-CoV2 infection.

Method To study single-cell B and T memory cells specific for the anti-SARS-CoV-2 response and characterize somatic mutations of immunoglobulin genes and TCR, in hospitalized and symptomatic patients and in patients cured of SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have recovered from CoV-2-SARS
* Adult patient (≥ 18 years old) with a positive SARS-CoV-2 PCR.
* Adult patient (≥ 18 years old) who has recovered from SARS-CoV-2 i.e. has been free of clinical symptoms for more than 15 days and has not been hospitalized and for less than 6 weeks.
* Patient affiliated to a social security scheme.

Patients hospitalized for SARS-CoV-2

* Adult patient (≥ 18 years old) with a positive SARS-CoV-2 PCR.
* Adult patient (≥ 18 years old) with clinical symptoms for more than 3 days and hospitalized.

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Patient under guardianship / curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Immunological memory: resolution of COVID-19 after SARS-CoV2 infection. | 5 years
  Biological blood collection: Blood samples taken in the course of the research will be part of a biological collection To study single-cell B and T memory cells specific for the anti-SARS-CoV-2 response and characterize somatic mutations of immunoglobulin genes and TCR, in hospitalized and symptomatic patients and in patients cured of SARS-CoV-2.

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Derived] Sokal A, Bastard P, Chappert P, Barba-Spaeth G, Fourati S, Vanderberghe A, Lagouge-Roussey P, Meyts I, Gervais A, Bouvier-Alias M, Azzaoui I, Fernandez I, de la Selle A, Zhang Q, Bizien L, Pellier I, Linglart A, Rothenbuhler A, Marcoux E, Anxionnat R, Cheikh N, Leger J, Amador-Borrero B, Fouyssac F, Menut V, Goffard JC, Storey C, Demily C, Mallebranche C, Troya J, Pujol A, Zins M, Tiberghien P, Gray PE, McNaughton P, Sullivan A, Peake J, Levy R, Languille L, Rodiguez-Gallego C, Boisson B, Gallien S, Neven B, Michel M, Godeau B, Abel L, Rey FA, Weill JC, Reynaud CA, Tangye SG, Casanova JL, Mahevas M. Human type I IFN deficiency does not impair B cell response to SARS-CoV-2 mRNA vaccination. J Exp Med. 2023 Jan 2;220(1):e20220258. doi: 10.1084/jem.20220258. Epub 2022 Nov 7. PMID 36342455
- [Derived] Attias P, Azzaoui I, El Karoui K, de La Selle A, Sokal A, Chappert P, Grimbert P, Fernandez I, Bouvier M, Samson C, Dahmane D, Rieu P, Nizard P, Fourati S, Sakhi H, Mahevas M; Mondor NephroCov Study Group. Immune Responses after a Third Dose of mRNA Vaccine Differ in Virus-Naive versus SARS-CoV-2- Recovered Dialysis Patients. Clin J Am Soc Nephrol. 2022 Jul;17(7):1008-1016. doi: 10.2215/CJN.00830122. Epub 2022 Jun 28. PMID 35764393